CLINICAL TRIAL: NCT00218153
Title: Naltrexone Augmentation of Nicotine Patch Therapy
Brief Title: Naltrexone Augmentation of Nicotine Patch Therapy - 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-13334-1; P50-13334-1
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2005-09

CONDITIONS: Tobacco Use Disorder
Keywords: nicotine dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Naltrexone

INTERVENTIONS:
Drug: Naltrexone

SUMMARY:
Naltrexone Augmentation of Nicotine Patch Therapy

DETAILED DESCRIPTION:
This double blind placebo controlled study is designed to determine whether naltrexone can be used to help reduce cigarette use and craving for cigarettes. Eligible participants will receive 21mg transdermal nicotine as an outpatient. In addition, participants will receive one of three doses of naltrexone (25,50 or 100mg) or a placebo and brief counseling over the course of six weeks with follow-up appointments three, six, and twelve months after the beginning of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and older
2. Willingness and ability to give written consent
3. Smoking 20 cigarettes per day for at least 1 year
4. At least one prior attempt to stop smoking
5. Baseline expired carbon-monoxide level of at least 10 ppm
6. Weigh at least 100 lbs.
7. English speaking
8. One person per household

Exclusion Criteria:

1. Pregnant or nursing women or women who do not use a reliable form of birth control
2. Unstable cardiac disease
3. History of dermatoses
4. Current alcohol dependence
5. Current use of opiates
6. A urine drug screen that is positive for opiates
7. Serious current neurologic, psychiatric or medical illness
8. Chronic pain conditions necessitating opioid treatment
9. Evidence of significant hepatocellular injury as evidence by SGOT or SGPT >3 x normal or elevated bilirubin
10. Current use of smokeless tobacco, pipes, cigars, nicotine gum or nicotine patch
11. Patients requiring concomitant therapy with any psychotropic drug or on any drug with a psychotropic component

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2000-11; Study Completion 2004-04

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie O'Malley, Ph.D., Principal Investigator — Substance Abuse Treatment Unit
Locations (2):
- United States (2):
  - Substance Abuse Treatment Unit, New Haven, Connecticut
  - VA Connecticut Health Care System, New Haven, Connecticut

REFERENCES:
- [Derived] King AC, Cao D, Zhang L, O'Malley SS. Naltrexone reduction of long-term smoking cessation weight gain in women but not men: a randomized controlled trial. Biol Psychiatry. 2013 May 1;73(9):924-30. doi: 10.1016/j.biopsych.2012.09.025. Epub 2012 Nov 22. PMID 23177384
- [Derived] O'Malley SS, Krishnan-Sarin S, McKee SA, Leeman RF, Cooney NL, Meandzija B, Wu R, Makuch RW. Dose-dependent reduction of hazardous alcohol use in a placebo-controlled trial of naltrexone for smoking cessation. Int J Neuropsychopharmacol. 2009 Jun;12(5):589-97. doi: 10.1017/S146114570800936X. Epub 2008 Sep 17. PMID 18796184